CLINICAL TRIAL: NCT04244526
Title: Distribution of Virulence Genes and Their Association With Clinical Presentation of Urinary Tract Infection and Antimicrobial Resistance Among Uropathogenic Escherichia Coli Isolated From Pregnant Women
Brief Title: Urinary Tract Infection in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NSHussein, Demonstrator of medical microbiology and immunology. Faculty of medicine. Assiut university, Assiut University
Other Study IDs: Urinary tract infection
Record Dates: First submitted 2020-01-25; First posted 2020-01-28 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group1: Group 1:pregnant women with cystitis
  Interventions: Other: Talking a urine sample
- Group2: Group 2: pregnant women with Pyelonephritis
  Interventions: Other: Talking a urine sample
- Group3: Group 3: pregnant women with asymptomatic bacteriuria
  Interventions: Other: Talking a urine sample

INTERVENTIONS:
Other: Talking a urine sample — Just taking a urine sample

SUMMARY:
* to describe the profile of uropathogenic E coli from Egyptian pregnant women with UTIs and a symptomatic bacteriuria.
* to determine the susceptibility pattern of our local isolated UPEC strains which is essential for optimal management of UTI.
* to evaluate the different virulence genes in UPEC isolates and their association with antibiotic resistance.
* to track common UPEC serogroups.
* to investigate the biofilm formation and the relationship between virulence genes and biofilm formation in UPEC strains isolated from patients.

DETAILED DESCRIPTION:
Urinary tract infection represents the most common bacterial infection in pregnancy and the third common cause of human infection after respiratory and intestinal infections. The infection can be life threatening and associated with serious complications. UTI can be associated with defined symptoms'symptomatic' or without symptoms 'asymptomatic'. Asymptomatic bacteriuria is defined as the presence of >100000 colony forming units/ml of urine of a single pathogen in two consecutive midstream clean catch urine specimen or on catheterization specimen from an individual without signs or symptoms associated with urinary or genital organs. Asymptomatic bacteriuria can lead to acute pyelonephritis in30%of pregnant women and complications such as early delivery, increase risk of hypertension, pre-eclampsia, low birth weight and postpartum endometritis. Ecoli accounts for most cases of symptomatic and asymptomatic bacteriuria in women, representing70 _90 %of the cases. The important virulence factors of uropathogenic ecoli can be broadly divided into two groups :bacterial cell surface factors and secreted factors. The emergence of drug resistant microorganism among Uropathogenic Escherichia coli strains increases the serious threat to global health. Ecoli often acquired genes coding for antibiotic resistance, beta-lactamase enzymes are the most frequent and play a key role, conferring resistance of bacteria to beta lactam antibiotic group such as penicillin and cephalosporins. Therefore, knowledge regarding local prevalence of uropathogenic ecoli and antimicrobial resistance is essential for optimal management of UTI.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who diagnosed through clinical examination and urine analysis. 3 groups : group 1 pregnant women with cystitis Group 2 pregnant women with Pyelonephritis Group 3 pregnant women with asymptomatic bacteriuria

Exclusion Criteria:

* pregnant women on antibiotics _Patients with any anatomical abnormalities in the urinary tract

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women at different trimesters with cystitis and pyelonephritis and asymptomatic bacteriuria
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of virulence genes in different isolated UPEC strains | Three months
  Measurment of virulence genes of Escherichia coli strains by molecular diagnosis as PCR technique to determine relationship between clinical presentation of urinary tract infection and distribution of virulence genes of strains

SECONDARY OUTCOMES:
Correlation between the virulence genes and antibiotic resistance | Seven months
  Measurment of virulence genes of escherichia coli strains by molecular diagnosis as PCR technique,and determine antibiotic susceptibility of ecoli strains between different groups of women to determine relationship between distribution of virulence genea and antibiotic susceptibility of strains